CLINICAL TRIAL: NCT01537679
Title: Meditation or Relaxation Used to Reduce Stress Response and Improve Cognitive Functioning in Older Family Dementia Caregivers
Brief Title: Meditation to Reduce Caregiver Stress
Acronym: Meditation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 10-000270; 09-03-086-01D
Record Dates: First submitted 2012-02-10; First posted 2012-02-23 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Depression NOS; Major Depressive Disorder; Anxiety NOS
Keywords: Caregiver; meditation; relaxation; stress
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Anxiety Disorders | interventions — Relaxation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Meditation Intervention (Other)
  Interventions: Behavioral: Kirtan Kriya meditation
- Relaxation Intervention (Other)
  Interventions: Behavioral: Relaxation

INTERVENTIONS:
Behavioral: Kirtan Kriya meditation — Meditation will be taught to 20 caregivers and supervised by Helen Lavretsky, M.D during their first visit. Meditation Kirtan Kriya will be performed for 12 minutes every day at the same time of the day for 8 weeks. Compliance will be monitored during visits and by daily diaries that will be reviewed at each visit.
  Other Names: Kundalini yoga meditation
  Arms: Meditation Intervention
Behavioral: Relaxation — Participants in the relaxation group will be asked to relax in a quiet place with eyes closed while listening to the music on the relaxation CD for 12 minutes every day at the same time for 8 weeks.
  Other Names: Relaxation techniques
  Arms: Relaxation Intervention

SUMMARY:
The purpose of this study is to determine whether meditation will reduce stress and depressive of adult caregivers of a person with dementia.

DETAILED DESCRIPTION:
This is an 8-week study to determine if meditation or listening to a relaxation CD will be effective in reducing depressive symptoms and stress, and in improving memory and cognition of caregivers who perform a daily meditation for 12 minutes a day for 8 weeks compared to caregivers listening to a relaxation CD for 12 minutes a day for 8 weeks. A second purpose of this study is to examine the role of genetic and inflammatory markers in response to listening to a relaxation CD and meditation.

ELIGIBILITY:
Inclusion Criteria:

1. Caregivers of relatives with dementia who present to the Alzheimer s Disease Center or other UCLA geriatric or memory clinics for evaluation of dementia, cognitive impairment and/or co-existing behavioral disturbances. Caregivers will be identified by the family member with dementia or the physician as the primary source of assistance and/or support, 45 years of age or older, in contact with the individual with dementia at least three times/week for no less than one year, and a relative of the care-recipient (i.e., spouse or adult child). This criteria will ensure that the caregivers had been affected by substantial chronic stress, and they will also meet criteria specified below.
2. Adequate written and oral fluency in English to understand and complete study forms and converse with study personnel.
3. Caregivers enrolled in the trial could meet the DSM-IVR criteria for minor depression or depression not otherwise specified (NOS), but not for other diagnosis of unipolar or bipolar major depression.
4. Score between 6 and 15 on the Hamilton Depression Rating Scale-24 item (HAM-D).
5. Score of 26 or higher on the Folstein Mini-Mental State Examination (MMSE).

Exclusion Criteria:

1. Current diagnosis of unipolar major depression, schizophrenia, bipolar, psychotic disorders including psychotic depression or dementia, attention deficit or hyperactivity disorder, anxiety, and alcohol or drug dependence. Those with lifetime history of psychiatric conditions other than unipolar major depression will be also excluded.
2. Medically unstable, delirious, or terminally ill (e.g. medical illness requiring hospitalization or intense outpatient management, such as heart disease; heart attack in the past 6 months; Congestive Heart failure; severe heart arrythmias; unstable hypertension; poorly controlled diabetes; recent head trauma with loss of consciousness; recent stroke with residual neurological symptoms; recent cancer with ongoing treatment, or any other medical conditions requiring weekly visits to PCP or pending surgery).
3. Level of suicidal risk precludes safe treatment on an outpatient basis with Hamilton Depression rating scale item number 3 rated as = 3.
4. Subjects reporting daily use of alcohol will be excluded.
5. Diagnosis of amnestic MCI by the analyses of delayed verbal recall on the California Verbal Learning Scale that will be 1.5 SD below the age/education adjusted norms for the general population.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-03; Primary Completion 2010-08 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (HDRS) | 8 weeks

SECONDARY OUTCOMES:
Caregiver Burden Scale | Week 1 and 8
Connor-Davidson Resilience scale (CD-RISC) | Week 1 and 8

CONTACTS AND LOCATIONS:
Overall Officials: Helen Lavretsky, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Semel Institute, Los Angeles, California, United States

REFERENCES:
- See also: Meditation to Reduce Caregiver Stress — http://www.semel.ucla.edu/latelife